CLINICAL TRIAL: NCT06316531
Title: A Randomized Controlled Phase III Clinical Study Comparing BL-M07D1 With T-DM1 in Patients With Unresectable Locally Advanced or Metastatic HER2-positive Breast Cancer
Brief Title: A Study Comparing BL-M07D1 With T-DM1 in Patients With Unresectable Locally Advanced or Metastatic HER2-positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-301
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1
- Control group (Experimental): Participants receive T-DM1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Experimental Group
Drug: T-DM1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Control group

SUMMARY:
This study is a registered phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-M07D1 in patients with unresectable locally advanced or metastatic HER2-positive breast cancer who had failed previous treatment with taxanes and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. No gender limit;
3. Age ≥18 years old and ≤75 years old at the time of signing the informed consent;
4. expected survival time ≥3 months;
5. Patients with histologically or cytologically confirmed, unresectable, locally advanced or metastatic HER2-positive breast cancer;
6. Provide the latest tumor tissues to the central laboratory for HER2 and HR detection;
7. Must have at least one measurable target lesion that meets the RECIST v1.1 definition;
8. ECOG 0 or 1;
9. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. Blood transfusion is not allowed within 14 days before the first use of the study drug, and no cell growth factor is allowed;
12. Coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT)≤1.5×ULN;
13. Urine protein ≤2+ or < 1000mg/24h;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 7 months after the end of treatment.

Exclusion Criteria:

1. Received chemotherapy with mitomycin C and nitrosourea within 6 weeks before the first dose, received surgery, chemotherapy, immunotherapy, etc. Within 4 weeks before the first dose, received endocrine therapy, palliative radiotherapy, and anti-tumor therapy approved by NMPA within 2 weeks before the first dose;
2. Previous use of HER2-ADC in the metastatic background;
3. Prior treatment with an ADC drug containing a camptothecin derivative (topoisomerase I inhibitor) as a toxin;
4. The history of severe cardiovascular and cerebrovascular diseases in the past six months was screened;
5. Complicated with pulmonary diseases leading to severe impairment of lung function;
6. History of ILD/interstitial pneumonia, current ILD/interstitial pneumonia, or suspected ILD/interstitial pneumonia; According to CTCAE v5.0 was defined as ≥ grade 3 pulmonary disease and ≥ grade 2 radiation pneumonitis;
7. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
8. Other primary malignancies diagnosed within 5 years before the first dose;
9. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
10. Patients with active central nervous system metastases;
11. Patients with a history of allergy to recombinant humanized antibody or to any of the excipents of BL-M07D1;
12. Patients with known hypersensitivity or delayed hypersensitivity to certain components of T-DM1 or similar drugs, or known contraindications to T-DM1;
13. History of autologous or allogeneic stem cell transplantation or organ transplantation;
14. Anthracycline-equivalent cumulative dose of adriamycin > 360 mg/m2;
15. Human immunodeficiency virus antibody positive, active hepatitis B virus infection, cirrhosis, or hepatitis C virus infection;
16. Serious infection within 4 weeks before the first dose of study drug; There was active pulmonary inflammation at the time of screening;
17. Patients with massive or symptomatic effusions or poorly controlled effusions;
18. Receiving active antiinflammatory drugs or any form of immunosuppressive therapy before randomization;
19. A history of severe neurological or psychiatric illness;
20. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
21. Intestinal obstruction, Crohn's disease, ulcerative colitis or chronic diarrhea;
22. Subjects who are scheduled to receive live vaccine or receive live vaccine within 28 days before the first dose;
23. Patients who were deemed by the investigator to be ineligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Herui Yao, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China